CLINICAL TRIAL: NCT01851213
Title: A Prospective Observational Study to Examine, in Routine Clinical Practice in the US, Practice Patterns and Impact on Clinical Decision Making Associated With the FoundationOne™ Next Generation Sequencing (NGS) Test
Brief Title: FoundationOne™ Test Registry Study
Acronym: FMI Registry
Status: Completed | Type: Observational
Sponsor: Foundation Medicine (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FMI-001-NGS-500
Record Dates: First submitted 2013-05-06; First posted 2013-05-10 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Cancer; Neoplasm Metastasis; Tumor
Keywords: genomics; cancer; registry; neoplasm metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FoundationOne™ Test Ordered: Patients for whom a FoundationOne™ test was ordered and a report is delivered.

SUMMARY:
This study is a prospective, multicenter, observational study to characterize utilization patterns of the FoundationOne™ test by oncologists under conditions of routine clinical practice in the US. The study will also examine impact of test results on subsequent clinical decisions regarding choice of therapy. The planned duration of the study is at least 2 years with 1 year for patient recruitment and a minimum 1-year follow-up period for each patient. Any patient for whom the treating physician has ordered a FoundationOne™ test and a report is delivered is eligible for participation on the study. Eligible patients from participating sites will be enrolled sequentially during the 1-year enrollment period. Sites will be required to maintain an enrollment log of all patients for whom the FoundationOne™ test has been ordered and document patient disposition and reasons for non-participation. All treatment decisions and clinical assessment will be made at the discretion of the treating physician per usual care and are not mandated by study design or protocol. Informed consent will be obtained from eligible patients prior to study entry.

DETAILED DESCRIPTION:
Molecular testing of tumors, using techniques such as next-generation sequencing (NGS), facilitates an individualized approach to cancer treatment by sub-classifying diseases on an individual basis. Physicians can utilize an in depth understanding of disease at a molecular level to optimize therapy by selecting the most appropriate drugs and therapeutic targets. Genomic profiling has identified multiple genomic aberrations that are predictive markers for treatment response with targeted therapeutics.

FoundationOne™ is a commercially available molecular diagnostics test, for all solid tumor types, that analyzes routine clinical specimens for somatic alterations in relevant cancer-related genes. This validated in vitro diagnostic test, is performed in a single Clinical Laboratory Improvement Amendments (CLIA) certified and College of American Pathologists (CAP) approved laboratory at Foundation Medicine, Inc. It provides individualized, potentially actionable information regarding a patient's molecular cancer subtype that can be used by physicians to tailor treatment options.

With the recent commercial availability of the FoundationOne™ test, knowledge gaps exist regarding practice patterns associated with the use of this test in routine clinical practice and the impact of this test on clinical decision making. There is limited information regarding physician and patient characteristics that determine which patients receive the test, rationale for patient selection, and how physicians interpret and use the test results. Findings from this study will help to optimize patient selection and maximize the clinical impact of the test in terms of guiding therapy.

ELIGIBILITY:
Inclusion Criteria:

The FoundationOne test was ordered by the treating physician under routine clinical practice

* Age ≥ 18 years
* Patient willing and able to provide informed consent
* Informed consent date is at least one day prior to the FoundationOne test report date

Exclusion Criteria:

There are no exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This Pilot Study will aim to enroll approximately 500 patients from a total of 40 oncology centers in the US over a 1-year time period. Any patient for whom the treating physician has ordered the FoundationOne test is eligible for inclusion in the study. In order to capture real-world treatment patterns, site recruitment will aim to include approximately 80% of sites (and 80% of patients) from the community oncology setting. Enrollment will be competitive and each site will be capped at a maximum of 15 patients.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2013-03; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Composite characterization of current real-world practice patterns in the use of the FoundationOne™ test and the effect of the FoundationOne™ test on clinical decision making across the US | Minimum 1 year follow-up
  Characterization of practice patterns for the use of the test described by:
  * Provider and site characteristics of patients receiving the FoundationOne test
  * Socio-demographic and clinical characteristics of patients receiving the FoundationOne test
  Examination of the effect of the test on clinical decision making by describing:
  * Subsequent treatment patterns for patients after receipt of test results
  * Clinician report outcomes regarding how test results guided clinical decision making

SECONDARY OUTCOMES:
Exploratory endpoints describing clinical outcomes in the study population | Minimum 1 year follow-up
  * Overall survival
  * 1-year survival
  * Overall progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Palmer, MD, Principal Investigator — Sr VP Medical Afairs
Locations (1):
- Evergreen Hematology/Oncology, Spokane, Washington, United States